CLINICAL TRIAL: NCT00346788
Title: The Subvastus Approach in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RL-001
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2008-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIS (Experimental): minimally invasive incision
  Interventions: Procedure: Surgical approach for total knee arthroplasty
- Standard (Active Comparator): Standard incision length
  Interventions: Procedure: Surgical approach for total knee arthroplasty

INTERVENTIONS:
Procedure: Surgical approach for total knee arthroplasty — total knee arthroplasty surgery using minimally invasive surgery or standard technique.

SUMMARY:
The purpose of this study is to determine if the observed benefits of minimally invasive total knee arthroplasty, namely decreased hospital stay and increased range of motion, can be achieved with standard knee arthroplasty using the subvastus approach.

ELIGIBILITY:
Inclusion Criteria:

* You are willing to take part in the study, including signing this form after carefully reading it.
* You are available for follow-up for a minimum of 24 months (2 years).
* You have no medical conditions that prevent you from having surgery.
* This is the primary (first) knee replacement for this knee
* You are fluent in English and are able to understand your responsibilities in this study.

Exclusion Criteria:

* Active, local or systemic infection
* Fibromyalgia or other chronic pain syndrome
* Inability to follow the study requirements
* Had this knee replaced before
* Had a previous surgery on this knee that would interfere with the MIS approach (examples are femoral-femoral bypass, femoral-popliteal bypass, and quadricepsplasty)
* Body Mass Index (BMI) > 35, as you would not be eligible for the MIS approach.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Post Operative
Range of motion at discharge and six weeks post-operatively | Discharge and six weeks post operative

SECONDARY OUTCOMES:
Wound complications | post operative until wound healed
Post-operative narcotic use | 24 months post operative
Post-operative blood loss | Post operative
The ability to straight-leg raise at two and twenty-four hours post-operatively | 2 and 24 hours post operative
Knee Society Clinical Rating Scale | pre-op, 6 months, 12 months, and 24 months post operative
SF-12 | pre-op, 6 months, 12 months, and 24 months post operative
WOMAC. | pre-op, 6 months, 12 months, and 24 months post operative

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD, FRCS(C), Principal Investigator — Capital Health, Canada
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada